CLINICAL TRIAL: NCT07171788
Title: Effects of Low Level Laser Therapy on Wrist Flexors Spasticity and Hand Functions in Patients With Stroke
Acronym: LLL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Hassan Amin Mohamed, principle investigator : heba hassan amin mohamed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005969
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: low level laser therapy; wrist flexor spasticity; hand function; stroke
MeSH Terms: conditions — Stroke | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: low level laser therapy and selected phyisical therapy program
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level laser therapy (Experimental): twenty patients will receive low level laser therapy three times a week for 6 weeks
  Interventions: Other: low level laser therapy; Other: selected physical therapy program
- selected physical therapy program (Active Comparator): twenty patients will recieve selected physical therapy program plus sham low level therapy three time a weeks for 6 weeks
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Other: low level laser therapy — patients will receive LLT. The LLLT system used in the study (ASA LASER M6) delivered 1.0 W in continuous wave at a wave length in the near infrared of 808 nm. The incident power density will be 670 mW/cm2.The probe head will held with light pressure in contact with the skin over the course of median nerve on the dysfunctional limb for 15 minutes. Protective goggles will be used to prevent direct eye contact of the laser beam. plus selected phyiscal therapy program
  Arms: low level laser therapy
Other: selected physical therapy program — patient will receive standard physical therapy program for wrist flexors spasticity post-stroke typically includes the following components: Passive stretching: Passive static or dynamic stretching of the wrist flexorss is the mainstay to reduce spasticity and Physical therapy exercises in form of specific techniques of proprioceptive facilitation, relaxation techniques, passive and self-passive motions, and proper limb positioning. plus sham low level laser therapy

SUMMARY:
this study will be conducted to investigate the effect of low level laser therapy (LLLT) on wrist flexors spasticity and hand functions in patient with stroke

DETAILED DESCRIPTION:
Spasticity is more often found in the flexors muscles of the upper limb (fingers, wrist, and elbow flexors) and extensor muscles of the lower limb (knee and ankle extensors). Wissel et al observed that spasticity developed most often in elbow (79%), wrist (66%), ankle (66%), and shoulder (58%).9 Lundstrom et al concluded that spasticity is observed more frequently in the upper extremities than in the lower extremities, and Urban et al found a higher degree of spasticity in the upper limb muscles. LLLT is thought to work through several mechanisms. Stimulating ATP production and increasing cellular energy. The therapy can cause vasodilation, improving circulation in the treated area. It may also reduce the production of inflammatory mediators and increase anti-inflammatory factors, while potentially stimulating the synthesis of growth-promoting factors that facilitate tissue healing, and renewal may be stimulated by this therapy. In the context of spasticity management, LLLT has garnered scientific interest as a possible intervention, although its efficacy remains under scrutiny .Hypothesized mechanisms of action include muscle tone reduction through enhanced circulation and decreased inflammation in muscular and adjacent tissues, potentially fostering the relaxation of hypertonic muscles. Certain research indicates that LLLT may modulate the release of neurotransmitters crucial to muscle contraction and relaxation processes.

ELIGIBILITY:
Inclusion Criteria:

* forty stroke patients with wrist flexors spasticity from both sex will be participate in this study
* Their age ranges from 45 to 60 years.
* Patients will be referred by neurological consultants.
* preserved cognitive system, i.e., ability to respond to verbal stimul
* Body mass index less than 30.
* Patients will be diagnosed by clinical and radiological examination.
* patients with wrist flexors spasticity according to modified ashworth scale score +1 to 2.

Exclusion Criteria:

* Patients with contractures, fractures, rigidity, and deformity
* Patients with cognitive impairments.
* Patients with visual, auditory impairment affecting their ability to complete tasks.
* Uncontrolled Diabetic patient.
* Presence of hypoesthesia and/or hyperesthesia of the involved upper limb.
* Other major neurological condition (e.g., Spinal cord injury, multiple sclerosis, Epilepsy, Meningitis, and Brain tumor).
* presence of neoplastic lesions at the site of application

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
spasticity | up to 6 weeks
  Modified ashworth scale will be used to assess spaticity according the following criteria,0: No increase in muscle tone
  1. Slight increase in muscle tone, with a catch and release or minimal resistance at the end of the range of motion when an affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested as a catch, followed by minimal resistance through the remainder (less than half) of the range of motion
  2. A marked increase in muscle tone throughout most of the range of motion, but affected part(s) are still easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
hand grip strength | up to 6 weeks
  hand held dynamometer will be used to assess hand grip strength
muscle stiffness | up to 6 weeks
  The MyotonPRO will be used to assess muscle stiffness. it is a new handheld device that conveniently assesses stiffness of muscles and tendons.the device effectively measures changes in muscle stiffness due to fatigue It is placed on the skin over the muscle. A brief, gentle tap from the probe causes the muscle to oscillate. The oscillations are analysed automatically by the device to calculate the muscle's mechanical characteristics, such as its tone, stiffness and how elastic it is.

SECONDARY OUTCOMES:
pain intensity | up to 6 weeks
  A visual analogue scale will be used to assess pain. This scale is used to assess the severity of pain. It consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero), to the worst pain (10) that the patient could feel.